CLINICAL TRIAL: NCT07057479
Title: Phase III, Adaptive, Multicenter, Randomized, Superiority, Double-Dummy, Double-Blind Clinical Trial to Evaluate the Efficacy and Safety of a Fixed-Dose Combination of a Sodium-Glucose Cotransporter-2 (SGLT2) Inhibitor and a Thiazolidinedione in the Treatment of Type 2 Diabetes Mellitus, Compared to Monotherapy, in Patients Treated With Metformin
Brief Title: Phase III Trial of SGLT2 Inhibitor and Thiazolidinedione Fixed-Dose Combination vs. Monotherapy in Type 2 Diabetes Patients on Metformin
Acronym: CONTROL
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic change in development priorities
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EF191
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Type 2 Diabetes Mellitus; T2DM; Fixed-dose combination; SGLT2 inhibitor; Thiazolidinedione; Dual therapy; Glycemic control; Insulin resistance; Randomized clinical trial; Phase III trial; Diabetes treatment; Oral antidiabetic drugs; Metformin adjunct therapy; HbA1c reduction; Cardiovascular risk factors; Renal protection; Diabetes complications; Monotherapy comparison; Drug combination efficacy; Diabetes management
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Diabetes Complications | interventions — 2,4-thiazolidinedione; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fixed-Dose Combination of SGLT2i /TZD + Metformin (Experimental): Participants receive a fixed-dose combination tablet containing two antidiabetic agents (an SGLT2 inhibitor and a thiazolidinedione) once daily, plus matching placebos for both comparator drugs to maintain blinding. All participants continue background metformin therapy (≥1000mg/day). Sample size: 136.
  Interventions: Drug: Fixed-dose combination of SGLT2 inhibitor and thiazolidinedione; Drug: Background Therapy (All Groups) - Metformin
- Control Group 1 - SGLT2 Inhibitor + Metformin (Active Comparator): Participants receive monotherapy with an SGLT2 inhibitor once daily, plus matching placebos for both the FDC and the thiazolidinedione comparator to maintain blinding. All participants continue background metformin therapy (≥1000mg/day). Sample size: 136.
  Interventions: Drug: Control Group 1 Intervention - SGLT2 inhibitor monotherapy; Drug: Background Therapy (All Groups) - Metformin
- Control Group 2 - Thiazolidinedione + Metformin (Active Comparator): Participants receive monotherapy with a thiazolidinedione once daily, plus matching placebos for both the FDC and the SGLT2 inhibitor comparator to maintain blinding. All participants continue background metformin therapy (≥1000mg/day). Sample size: 136.
  Interventions: Drug: Control Group 2 Intervention - Thiazolidinedione monotherapy; Drug: Background Therapy (All Groups) - Metformin

INTERVENTIONS:
Drug: Fixed-dose combination of SGLT2 inhibitor and thiazolidinedione — Oral fixed-dose combination tablet containing an SGLT2 inhibitor and a thiazolidinedione, administered once daily. Participants also receive matching placebos for both comparator drugs to maintain blinding. All participants continue background metformin therapy (≥1000mg/day).
  Arms: Fixed-Dose Combination of SGLT2i /TZD + Metformin
Drug: Control Group 1 Intervention - SGLT2 inhibitor monotherapy — Oral tablet containing an SGLT2 inhibitor, administered once daily. Participants also receive matching placebos for both the fixed-dose combination and the thiazolidinedione comparator to maintain blinding. All participants continue background metformin therapy (≥1000mg/day). This represents standard monotherapy for comparison against the combination approach.
  Arms: Control Group 1 - SGLT2 Inhibitor + Metformin
Drug: Control Group 2 Intervention - Thiazolidinedione monotherapy — Oral tablet containing a thiazolidinedione, administered once daily. Participants also receive matching placebos for both the fixed-dose combination and the SGLT2 inhibitor comparator to maintain blinding. All participants continue background metformin therapy (≥1000mg/day). This represents standard monotherapy for comparison against the combination approach.
  Arms: Control Group 2 - Thiazolidinedione + Metformin
Drug: Background Therapy (All Groups) - Metformin — Extended-release metformin tablets (≥1000mg daily) continued as background therapy for all participants throughout the study duration.

SUMMARY:
This clinical trial is studying whether combining two commonly used diabetes medications into a single pill works better than taking them separately for people with type 2 diabetes who are already on metformin. Both medications work in different ways to lower blood sugar - one helps remove excess sugar through urine while the other helps the body use insulin better.

The study has two main goals:

To see if the combined pill controls blood sugar more effectively than either medication alone

To check if combining them reduces common side effects like weight gain and swelling that can occur with one of the medications

Participants will be randomly assigned to one of three groups:

The new combination pill

One of the standard diabetes medications alone

The other standard diabetes medication alone

All participants will take their assigned treatment daily and attend regular clinic visits for monitoring. Doctors will track blood sugar control, weight changes, and any side effects throughout the study period.

This research could lead to a simpler treatment option that combines the benefits of both medications while potentially minimizing side effects. For people with diabetes who often need multiple medications, a combined pill might make treatment easier to manage while providing better blood sugar control.

DETAILED DESCRIPTION:
This phase III clinical trial investigates a fixed-dose combination (FDC) of two established antidiabetic medications with complementary mechanisms of action: an SGLT2 inhibitor and a thiazolidinedione (TZD). The study aims to evaluate whether combining these medications in a single tablet provides superior glycemic control compared to either medication alone in patients with type 2 diabetes who are already on metformin therapy.

The SGLT2 inhibitor component lowers blood glucose by increasing urinary glucose excretion, while the TZD component improves insulin sensitivity. Previous studies have shown that these drug classes may offer complementary benefits for metabolic control and cardiovascular risk reduction. However, the TZD component has been associated with side effects including fluid retention and weight gain in some patients. This trial will assess whether the combination can maintain the therapeutic benefits of both drugs while potentially reducing TZD-related adverse effects.

The randomized, double-blind, double-dummy design compares three treatment arms: the FDC, SGLT2 inhibitor monotherapy, and TZD monotherapy. The primary endpoint is the change in HbA1c from baseline after 24 weeks of treatment. Secondary endpoints include measures of safety, tolerability, and additional metabolic parameters.

Participants will undergo regular monitoring including blood tests, physical examinations, and safety assessments throughout the study period. The trial includes specific protocols for detecting and managing potential side effects, particularly those related to fluid retention.

This study addresses an important clinical question regarding optimal treatment strategies for type 2 diabetes, particularly the potential advantages of fixed-dose combinations in simplifying treatment regimens while maintaining efficacy and safety. The results may provide evidence for a new therapeutic option that combines the established benefits of these two drug classes while potentially mitigating some limitations of monotherapy approaches.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age ≥18 years
* Diagnosis of type 2 diabetes (T2DM)
* HbA1c 7.5-10% while on stable metformin monotherapy (≥1000 mg/day) for ≥12 weeks
* ≥80% adherence to run-in medication

Exclusion Criteria:

* Type 1 diabetes or other specific diabetes types (e.g., monogenic, pancreatic, or drug-induced)
* Severe hyperglycemia (≥270 mg/dL) or diabetic ketoacidosis in past 12 weeks
* Hypersensitivity to study drugs or excipients
* Pregnancy, lactation, or planning pregnancy
* Severe diabetic complications (proliferative retinopathy, severe neuropathy)
* Major cardiovascular events in past 12 weeks (e.g., myocardial infarction, heart failure NYHA III/IV)
* Uncontrolled hypertension (SBP >180 mmHg or DBP >110 mmHg)
* Moderate/severe renal impairment (eGFR <45 mL/min/1.73m²)
* Liver disease (cirrhosis, active hepatitis)
* History of malignancy (except treated skin cancers) in past 5 years
* Use of non-metformin antidiabetics or weight-loss drugs in past 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-09 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Change in glycated hemoglobin (HbA1c) from baseline to week 24 | From baseline to week 24

SECONDARY OUTCOMES:
Proportion of participants achieving HbA1c <7.0% at week 24 | At week 24
Change in fasting plasma glucose from baseline to week 24 | Baseline to week 24
Incidence of adverse events (AEs) over 24 weeks | Baseline to week 24
Incidence of peripheral edema over 24 weeks | Baseline to week 24
Incidence of moderate/severe hypoglycemia (Level 2/3) over 24 weeks | Baseline to week 24

OTHER OUTCOMES:
Change in body weight from baseline to week 24 | Baseline to week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofarma Laboratórios S.A, Itapevi, São Paulo, Brazil